CLINICAL TRIAL: NCT05421130
Title: Clinical Investigation of Clinical Safety and Performance of the SP-GRIPFLOW, Selective Cerebral Perfusion Catheter When Used for Cerebral Perfusion During Aortic Arch Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fuji Systems Corporation (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL73323.100.21
Record Dates: First submitted 2022-04-22; First posted 2022-06-16 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Aortic Aneurysm; Aortic Dissection; Aortic Arch Aneurysm; Aortic Arch; Aneurysm, Dissecting
MeSH Terms: conditions — Aortic Aneurysm; Aortic Dissection; Aneurysm, Aortic Arch; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SP-GRIPFLOW (Other): This is a single-arm clinical investigation. Enrolled subjects will have cerebral perfusion with the investigational device during surgical repair of the aortic arch. A total of 1-3 investigational devices will be used per subject.
  Interventions: Device: Selective Cerebral Perfusion Catheter

INTERVENTIONS:
Device: Selective Cerebral Perfusion Catheter — This product is intended to be placed in the branches of the aortic arch for the cerebral perfusion during surgery of aorta.
  Other Names: SP-GRIPFLOW

SUMMARY:
The purpose of this study is to determine if the SP-GRIPFLOW catheter (the catheter designed by Fuji Systems) is safe and how well it functions. The information from this research will be used to help decide if the device should be approved for sale in the European Union. The SP-GRIPFLOW catheter may not yet be used by investigators outside of the study.

Through the study, FUJI will prove that the target flow as measured by the flow through the catheter(s)(cumulative flow for multiple catheters) was confirmed in 95% of cases.

DETAILED DESCRIPTION:
The SP-GRIPFLOW catheter is a catheter that is used to transport blood from the aortic arch to your brain during surgery on the aorta. The procedure in which the catheter is used does not differ from the procedure as performed with current catheters. Furthermore, the SP-GRIPFLOW catheter is used in a similar manner as other catheters that are currently on the market. Contrary to available catheters, the SP-GRIPFLOW has a ribbed surface on the balloon end of the device, which aims to improve the grip of the balloon in order to reduce chances of dislocation from the target artery.

Clinical trials are needed to obtain or expand knowledge about the safety, suitability and effi-cacy of medical devices. This is why the legislative authority has specified in the law on medi-cal devices that new medical devices must be clinically tested. The clinical trial that we present to you here was - as required by law - granted a favourable opinion by an ethics committee and approved by the competent authority. This clinical trial will be conducted at up to 5 sites in the European Union; a total of approximately 149 persons will participate in it. The study is being initiated, organised, and financed by Fuji Systems Corporation, the sponsor of this study.

ELIGIBILITY:
Inclusion Criteria:

Subjects shall fulfil all of the following criteria:

* Is willing and able to understand and sign informed consent, and has signed an information and inform consent
* Is male or female
* Is minimum 18 years of age when signing the informed consent
* Has been diagnosed with an aortic arch aneurysm or chronic dissection with an indication for open arch repair
* Is indicated for elective open/hybrid aortic arch repair with cerebral perfusion
* Is willing and able to comply to the schedule of assessment of the clinical investigation
* Has a target vessel diameter appropriate for the use of the SPGRIPFLOW Catheter (12Fr, 14Fr or16Fr)

Exclusion Criteria:

Subjects shall fulfil none of the following criteria:

* Aortic dissection or rupture which requires acute surgery
* Emergency surgery
* American Society of Anesthesiologists (ASA) Class >IV
* Is currently participating in, or has recently exited from (within 30 days prior to screening for this clinical investigation), or plans to be enrolled (during the course of this clinical investigation) in another clinical investigation that may affect the endpoints of this clinical investigation.
* Had cerebral perfusion with another similar device/competitor device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
"Successful perfusion" defined by flow rate through the catheter (mL/kg/min) | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  The primary endpoint is defined by blood flow through the SPGRIPFLOW and perfusion of the brain during open surgical repair of the distal aortic arch. Blood flow (and perfusion) is assessed by the flow rate through the cannula(s) compared to the target flow rate. Successful perfusion is defined when the flow rate through the catheter(s) equals the target flow rate (mL/kg/min). The perfusion flow rate will be monitored throughout the procedure. The target flow rate will be preoperatively defined by the investigator

SECONDARY OUTCOMES:
"Adequate flow rate" assessed by a clinically relevant through the catheter(mean and maximum flow rate「mL/kg/min」). endpoints | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  The secondary endpoint of this study will focus on assessment of adequate flow rate through the SP-GRIPFLOW. Whether the SPGRIPFLOW allows for an adequate flow rate will be assessed by a clinically relevant flow through the catheter(s) (mean and maximum flow rate). A clinically relevant perfusion flow rate of 10-15 mL/min/kg was defined from scientific literature.

OTHER OUTCOMES:
The nature, severity and incidence of adverse events at 30-days post-procedure | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  The safety of the SP-GRIPFLOW Catheter will be assessed by the nature, severity and incidence of adverse events at 30-days post-procedure. The adverse events found for the SP-GRIPFLOW will be compared to the current knowledge and state of the art to assess whether the device is associated with acceptable safety outcomes. No formal hypothesis testing will be performed for the safety endpoint of this clinical investigation.
The collection of an intraoperative parameters(Number of catheter dislocations from target artery (Units)) | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  Number(Units) of catheter dislocations from target artery will be assessed as exploratory endpoints.
The collection of an intraoperative parameters(Near-infrared spectroscopy (O2 saturation)) | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  Near-infrared spectroscopy (O2 saturation) will be assessed as exploratory endpoints.
The collection of an intraoperative parameters (Perfusion pressure (mmHg)) | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  Perfusion pressure (mmHg) will be assessed as exploratory endpoints. Perfusion pressure is interpreted as below items. Line pressure Pressure at the tip of SP-GRIPFLOW (if available) Radial blood pressure, left and right
The collection of an intraoperative parameters (Circulatory arrest time (minutes)) | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  Circulatory arrest time(minutes) will be assessed as exploratory endpoints.
The collection of an intraoperative parameters (Selective cerebral perfusion time (minutes)) | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  Selective cerebral perfusion time (minutes) will be assessed as exploratory endpoints.
The collection of an intraoperative parameters(Perfusion flow rate (mL/kg/min) (maximum and minimum)) | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  Perfusion flow rate (mL/kg/min) (maximum and minimum) will be assessed as exploratory endpoints.
The collection of an intraoperative parameters(Degree of hypothermia (degrees Celsius)) | The enrolment period is expected to take approximately 15 months. The duration of the subject's participation is circa 1 month. The total expected duration of the clinical investigation is, therefore, approximately 16 months.
  Degree of hypothermia (degrees Celsius) will be assessed as exploratory endpoints.
  (tympanic membrane or nasal temperature [for cerebral perfusion temperature measurement] and any of followings if available: rectal temperature, bladder temperature, or esophageal temperature [for systemic circulation temperature measurement])

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (3):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Campus Freiburg: Hugstetter Straße 55
  - Universitätsklinikum Frankfurt, Frankfurt, Theodor-Stern-Kai 7,
  - Herzzentrum Leipzig GmbH, Leipzig, Universitätsklinik Für Herzchirurgie Strümpellstraße 39
- Netherlands (2):
  - St.Antonius Hospital, Nieuwegein, Koekoekslaan 1, 3435 CN
  - Radboud universitair medisch centrum, Nijmegen

IPD SHARING:
Plan to Share IPD: No